CLINICAL TRIAL: NCT05264103
Title: Assessment of Robotic Assistance on Gait Parameters.
Brief Title: Assessment of Robotic Assistance on Gait Parameters Among Healthy Subjects and Brain Damaged Patients
Acronym: MARAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/4OCT/404
Record Dates: First submitted 2021-12-22; First posted 2022-03-03 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group. (Experimental): Healthy subjects and brain damaged patients with gait disorder.
  Interventions: Device: Exoskeleton for gait rehabilitation (Atalante)

INTERVENTIONS:
Device: Exoskeleton for gait rehabilitation (Atalante) — Subjects will walk with different levels of assistance given by the robot.

SUMMARY:
The main objective of this study is to quantitatively assess the robotic assistance given by an exoskeleton on patients gait parameters. Patients will be asked to walk with- and without the exoskeleton on a treadmill. During the study, the biomechanical and the energy consumption will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis due to stroke
* Min 18 years
* Time since stroke > 15 days
* Ability to understand instructions
* Ability to do gait analysis on the treadmill

Exclusion Criteria:

- Contraindication for the use of the robot Atalante

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Energy cost (J.kg/m) | 1 week
  A nasal mask is fitted to the subject to measure oxygen consumption (VO2) and carbon dioxide production (VCO2). The ratio between VCO2 and VO2 is used to calculate the respiratory exchange ratio (RER). The Joules of energy expended per liter of oxygen consumed were computed depending on the RER. RER is assessed in a standing and walking condition. Finally, the energy cost is obtained by the ratio "walking expended minus standing'' divided by speed.

SECONDARY OUTCOMES:
Temporo-spatial parameters of gait: step length | 1 week
  Reflective landmarks positioned on precise anatomic sites were used to compute spatiotemporal variables. 8 infra-red camera are used to asess step length (m).
Temporo-spatial parameters of gait: stance phase | 1 week
  Reflective landmarks positioned on precise anatomic sites were used to compute spatiotemporal variables. 8 infra-red camera are used to assess stance phase (%).
Temporo-spatial parameters of gait: cadence | 1 week
  Reflective landmarks positioned on precise anatomic sites were used to compute spatiotemporal variables. 8 infra-red camera are used to assess cadence (step/min).
Segmental kinematics of gait (°) | 1 week
  Reflective landmarks positioned on precise anatomic sites were used to compute kinematic variables. Data from landmarks are collected with 8 infra-red camera. From Euler angles, it allowed the computation of angular displacements of the pelvis, hip, knee and ankle in the three planes of space.
Muscle activation | 1 week
  Electrodes are placed on different muscles to record muscles activity.
Mechanical work (J.kg/m) | 1 week
  The total positive mechanical work performed by the muscles during gait is calculated by the sum of external work (performed to move the body center of mass) and internal work (performed to move the body segments relative to the body center of mass)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lejeune, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium